CLINICAL TRIAL: NCT01044602
Title: Metabolic Surgery vs. Medical Management for Resolution of Type II Diabetes: A Prospective Group Match Study
Brief Title: Metabolic Surgery Versus Medical Management for Resolution of Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Bradley MD (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor-Investigator, David Bradley MD, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009H0282; MS vs. MM for DM2 (Other: Dept identifier)
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Obesity; Type 2 Diabetes Mellitus; Roux-en-Y Gastric Bypass Surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best Medical Management (Active Comparator): Patients elect to treat obesity and type 2 diabetes mellitus through best medical management.
  Interventions: Other: Laboratory evaluations, sleep study; Other: Best Medical Management
- Surgical Treatment (Active Comparator): Patients with type 2 diabetes mellitus choice to treat obesity with Roux-en-Y gastric bypass.
  Interventions: Other: Laboratory evaluations, sleep study; Procedure: Roux-en-Y gastric bypass surgery

INTERVENTIONS:
Other: Laboratory evaluations, sleep study — Fasting plasma glucose, liver function tests, chem-7, HOMA-IR, HBA1C, lipid profile, indirect calorimetry.
Other: Best Medical Management — Standard of care.
  Arms: Best Medical Management
Procedure: Roux-en-Y gastric bypass surgery — Surgical treatment.
  Arms: Surgical Treatment

SUMMARY:
Best medical management and gastric bypass surgery is a way to treat diabetes as part of regular medical care (standard of care). However, gastric bypass surgery is not a way to treat diabetes as part of regular medical care (standard of care).

DETAILED DESCRIPTION:
Best medical management and gastric bypass surgery are ways to treat obesity as part of regular medical care (standard of care). Best medical management is a way to treat diabetes as part of regular medical care (standard of care). However, gastric bypass surgery is not a way to treat diabetes as part of regular medical care (standard of care). But, studies suggest that diabetes gets better or goes away after gastric bypass surgery. This study is being done to find out if diabetes gets better or goes away completely after a patient has gastric bypass surgery as part of regular medical care (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 70
* BMI 35 or greater
* HbA1c>6.5%
* Stable weight
* Stable medications

Exclusion Criteria:

* Coagulopathy
* Liver cirrhosis
* C-peptide <1 ng/ml (off insulin)
* Diagnosis of severe eating disorder
* Untreated endocrine disorder
* Use of medication for weight loss in the past 6 months
* Use of medication for weight loss in the last 6 months (with the exception of orlistat)
* Pregnancy
* Coagulopathy
* Liver cirrhosis
* Incurable, malignant, or debilitating disease
* Severe eating disorder
* Use of weight loss medication in the last 6 months, with the exception of orlistat
* Untreated endocrine disorder
* Pregnant
* Inability to provide informed consent

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Resolution of type 2 diabetes mellitus, determined by oral glucose tolerance test. | 2 years
Resolution of obesity co-morbidities including hypertension, OSA, and hyperlipidemia | 2 years

SECONDARY OUTCOMES:
Improvement in glucose control | 2 years
Improvement in control of chronic co-morbidities | 2 years
Identify predictors of success with regard to improved co-morbidities and velocity of weight loss | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Asem Ali, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States